CLINICAL TRIAL: NCT05402878
Title: RECANALISATION THERAPY IN ISCHEMIC STROKE DUE TO BASILAR ARTERY OCCLUSION IN PEOPLE 115 HOSPITAL, VIETNAM
Brief Title: OUTCOME AND SAFETY OF RECANALIZATION TREATMENTS IN ISCHEMIC STROKE DUE TO ACUTE BASILAR ARTERY OCCLUSION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: 115 People's Hospital (Other Government)
Responsible Party: Principal Investigator, NGUYEN THI BICH HUONG, Investigator, 115 People's Hospital
Other Study IDs: People 115 Hospital
Record Dates: First submitted 2022-05-26; First posted 2022-06-02 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Basilar Artery Occlusion
Keywords: BASILAR ARTERY OCCLUSION; RECANALISATION THERAPY

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: Recently, two prospective multicenter RCT reported a potential beneficial effect of endovascular thrombectomy (EVT) in patients with an acute symptomatic basilar artery occlusion (BAO). However, the high rate of crossover in BEST study and the long-term of recruitment in BASICS study influenced the validity of the results.

Objective: To assess the outcomes and prognostic factors of recanalization therapy in patients with BAO, caused by a CTA/MRA/DSA confirmed occlusion of the basilar artery.

Study design: This is a prospective observational study. Study population: Patients with acute ischemic stroke and a confirmed basilar artery occlusion by CTA/MRA/DSA.

Main study parameters/outcomes: Favorable outcome at day 90 defined as a modified Rankin Score (mRS - functional scale) of 0-3. The estimate will be adjusted for the known prognostic variables age, time from onset to treatment, stroke severity (NIHSS), PC ASPECT and collateral flow and adjusted and unadjusted estimates with corresponding 95% confidence intervals will be reported.

DETAILED DESCRIPTION:
Acute basilar artery thrombosis is associated with a poor prognosis. Prevalence of basilar artery occlusion are not known in Vietnam.Various treatments were tried in groups of patients with acute ischemic stroke due to basilar artery occlusion, but evidence based was not cleared previous studies. Therefore, we conduct this study to evaluate the efficacy and safety of recanalization therapies, which included intravenous thrombosis alone, endovascular alone, or bridging IVT and endovascular, in basilar artery occlusion stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms and signs compatible with ischemia in the basilar artery territory.
* Basilar artery occlusion (BAO) confirmed by CTA or MRA or DSA.
* Age 18 years or older
* Patients were treated with one of these among therapies IVT alone, bridging IVT and thrombectomy or thrombectomy alone..

Exclusion Criteria:

* Patients did not agree to enroll.

Imaging exclusion criteria:

* High-density lesion consistent with hemorrhage of any degree
* Significant cerebellar mass effect or acute hydrocephalus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were acute ischemic stroke due to basilar artery occlusion admitted People 115 Hospital and treated recanalisation therapies : intravenous tPA, bridging tPA and thrombectomy or thrombectomy alone.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
favourable outcome | 90 (± 14 days) after procedure
  a modified Rankin Score of 0-3

SECONDARY OUTCOMES:
good outcome | 90 (± 14 days) after procedure
  a modified Rankin Score of 0-2
mortality | 90 (± 14 days) after procedure
  Number of subjects who died at 90-day follow-up/total number of subjects who participated in 90-day follow-up) x100%.
Dichotomized mRS score | 90 (± 14 days) after procedure
  mRS (0-2 versus 3-6 and 0-4 versus 5-6 )
Symptomatic intracerebral hemorrhage (sICH) | within 72 hours after procedure
  SICH means any hemorrhage with neurological deterioration, as indicated by an NIHSS score that was higher by ≥4 points than the value at baseline or the lowest value in the first 72 hours or any hemorrhage leading to death.
Any intracerebral hemorrhage | within 72 hours after procedure
  intracerebral hemorrhage was defined according ECASS definition.
Procedural related complications | Perioperative period
  arterial perforation, arterial dissection, embolization in a previously uninvolved vascular territory and so on

CONTACTS AND LOCATIONS:
Overall Officials: Huy Thang Nguyen, Professor, Study Director — People 115 Hospital
Locations (1):
- People 115 Hospital, Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided